CLINICAL TRIAL: NCT02848469
Title: Randomized Control Trial of Omega-3 Fatty Acids Compared to Placebo in the Prevention of Psychosis in Very High Risk Individuals
Brief Title: Irish Omega-3 Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Damian O'Driscoll, Academic Study Coordinator, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMRI 11T-011
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders | interventions — Eicosapentaenoic Acid; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 fatty acids (Active Comparator): Subjects will receive food supplements in the form of 200ml juice drinks, containing either the active component, 1000mg of eicosapentaenoic acid and 1000mg docosahexaenoic acid, or matching placebo for a duration of six months. Neither the active nor the placebo food supplements taste of fish, so the subject will be blind to whether he/she is receiving the active intervention or placebo.
  Interventions: Dietary Supplement: 1000mg of eicosapentaenoic acid and 1000mg docosahexaenoic acid
- placebo 200ml juice drinks (Placebo Comparator): 200ml juice drinks
  Interventions: Dietary Supplement: 1000mg of eicosapentaenoic acid and 1000mg docosahexaenoic acid

INTERVENTIONS:
Dietary Supplement: 1000mg of eicosapentaenoic acid and 1000mg docosahexaenoic acid

SUMMARY:
The Irish Omega-3 study is a clinical trial designed to investigate the potential of Omega-3 fatty acids in the reduction of risk of psychosis.

The study is being coordinated by the HRB Clinical Research Facility at University College Cork. The Principal Investigator is Dr Maeve Rooney, Consultant Psychiatrist in the Mercy University Hospital, Cork. The study will be carried out in collaboration with the HRB Clinical Research Facility in Dublin in prior to rolling out to other centres around Ireland.

The Study is funded by Stanley Medical Research Institute, a non-profit organization supporting research on the causes of, and treatments for, schizophrenia and bipolar disorder. It is the largest provider of funding for research in serious mental illness outside of the U.S. government.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be aged between 13 and 50 years.
* Written informed consent will be obtained from subjects, or, in the case of those under - eighteen, from their parent or guardian, with the assent of the participant.
* Subjects meet the criteria of UHR, according to the Structured Interview for Prodromal Syndromes (SIPS) (Cannon et al., 2008, Woods et al., 2009).

Exclusion Criteria:

* Previous psychotic episode of at least one week's duration.
* Previous manic episode of at least one week's duration.
* Acute suicidal or aggressive behaviour.
* Substance dependence.
* Lactose intolerance/Milk allergy
* Intellectual disability, which in the opinion of the investigator would affect the person's ability to participate in the trial.
* Previous treatment with an antipsychotic or mood stabiliser for a psychiatric indication longer than 2 weeks in the previous three months.
* Consumption of over the counter or prescribed omega-3 fatty acids supplements within 12 weeks of entering the trial.
* Pregnancy/breast-feeding.
* Severe inter-current illness that may affect the ability of the participant to take part in the trial.

Ages: 13 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-09; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
To ascertain the effectiveness of Omega-3 fatty acid supplements in reducing transition to psychosis in individuals who are at ultra high risk of developing psychosis. | Assessments at baseline, 12 weeks, 24 weeks and 52 weeks
  The primary endpoint will be transition to psychosis, as determined by the Structured Interview for Psychosis-Risk Syndromes (SIPS).

SECONDARY OUTCOMES:
2. To assess in a subgroup of subjects the association of fatty acid changes, that is the blood Omega-3 to Omega-6 ratio, with the primary outcome. | Samples taken at baseline and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Facility, Cork, Ireland